CLINICAL TRIAL: NCT01317082
Title: Use of the Pressure Right Device After Laparoscopic Surgery
Status: No longer available | Type: Expanded Access
Sponsor: Therapeutics: 101 Inc. (Industry)
Responsible Party: Paul White, Ph.D, M.D., White Mountain Institute
Other Study IDs: JDL20-11
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-02

CONDITIONS: Nausea; Vomiting
Keywords: Postoperative Nausea & Vomiting.
MeSH Terms: conditions — Nausea; Vomiting; Postoperative Nausea and Vomiting | interventions — Acupressure

INTERVENTIONS:
Device: Acupressure — P 6 Pressure Point
  Other Names: Pressure Right

SUMMARY:
The primary objective is to test the hypothesis that the use of the Pressure Right device in combination with ondansetron and dexamethasone would result in a lower incidence of postoperative vomiting (emesis) than the combination of antiemetic therapy alone.

DETAILED DESCRIPTION:
The study design is a randomized, double-blinded and sham-controlled evaluation of the adjunctive Acupressure on the P6 point with Pressure Right to reduce the incidence of PONV and the need for rescue antiemetics leading to an improve quality of recovery after laparoscopic and ENT surgery. The two proposed study groups are: Group 1 (Sham-Control) 50 patients, will receive the sham Pressure Right (without acupressure button)30-45 min before induction of anesthesia and will be kept in place for 24h after discharge, and Group 2 (Pressure Right) 50 patients, will receive the Pressure Right device 30-45 min before induction of anesthesia and will be kept in place for 24h after discharge. In addition, all 100 study patients will receive a combination of antiemetics (ondansetron and dexamethasone) during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo major laparoscopic and ENT surgery procedures under genertal anesthesia.
* ASA Class I-III adults of either sex
* Willingness and ability to sign an informed consent document.

Exclusion Criteria:

* Patients with known allergy, hypersensitivity or contraindications to 5-HT3 antagonist.
* Patients experienced vomiting or retching within 24 h before surgery.
* Patients with clinically-significant medical conditions.
* Pregnant and lactating women.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult